CLINICAL TRIAL: NCT00151424
Title: A Multicenter, Randomized, Double-Blind, Flexible-Dose, 6-Week Trial of the Efficacy and Safety of Asenapine Compared With Placebo Using Olanzapine Positive Control in Subjects With an Acute Exacerbation of Schizophrenia
Brief Title: Efficacy and Safety of Asenapine With Placebo and Olanzapine (41022)(P05947)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05947; Hera; 41022
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — asenapine; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): asenapine 5-10mg BID
  Interventions: Drug: asenapine
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 3 (Active Comparator): olanzapine 10-20 mg QD
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: asenapine — Asenapine 5-10mgBID
  Arms: 1
Drug: Placebo — Matched against asenapine and olanzapine
  Arms: 2
Drug: Olanzapine — 10-20 mg QD
  Arms: 3

SUMMARY:
Schizophrenia is a brain disease. The primary features of schizophrenia are characterized by Positive symptoms (symptoms that should not be there, inability to think clearly, to distinguish reality from fantasy i.e., hearing voices) and Negative symptoms (a reduction or absence of normal behaviors or emotions, i.e., unable to manage emotions, make decisions and relate to others). Other symptoms include reduced ability to recall and learn new information, difficulty with problem solving, or maintaining productive employment. The symptoms of schizophrenia may be due to an imbalance in chemicals in the brain, primarily dopamine and serotonin, which enables brain cells to communicate with each other.

Asenapine is an investigational drug that may help to correct the imbalance in dopamine and serotonin. This is a 6 week study to test the efficacy and safety of asenapine and a comparator agent (olanzapine) in the treatment of patients with schizophrenia. Patients that complete this trial will have the option of continuing in an additional one year extension trial.

ELIGIBILITY:
Inclusion Criteria:

* Currently suffering from an acute exacerbation of schizophrenia.

Exclusion Criteria:

* Have an uncontrolled, unstable medical condition. Have any other psychiatric disorder other than schizophrenia as a primary diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2005-02-15 (Actual); Primary Completion 2006-01-06 (Actual); Study Completion 2006-02-06 (Actual)

PRIMARY OUTCOMES:
Change in total Positive and Negative Syndrome Scale (PANSS) score at endpoint (6-week double-blind or last assessment after baseline) from baseline | Screen, baseline, days 4, 7, 14, 21, 28, 35, 42
  A 30-item, clinician rated instrument for assessing the symptoms of schizophrenia. Ratings for each item could range from 1 (absent) to 7 (extreme).

SECONDARY OUTCOMES:
Changes in PANSS subscale and Marder factor score Clinical Global Impression-Severity of Illness (CGI-S) scores | Screen, baseline, Days 4,7,14,21,28,35,42
  This was not a prespecified key secondary outcome
Clinical Global Impression Improvement (CGI-I) scores | Days 4,7,14,21,28,35,42
  This was not a prespecified key secondary outcome
Neurocognition and cognitive functioning | Baseline , day 42
  This was not a prespecified key secondary outcome
Anxiety | Baseline, day 42
  This was not a prespecified key secondary outcome
Suicidal thinking | Baseline, day 42
  This was not a prespecified key secondary outcome
Quality of life and patient functionality | Baseline, day 42
  This was not a prespecified key secondary outcome
Readiness to discharge, at scheduled assessments and endpoint from baseline | Baseline up to day 14
  This was not a prespecified key secondary outcome
Extrapyramidal symptoms | Baseline, Days 4,7,14,21,28,35,42
  This was not a prespecified key secondary outcome
Laboratory parameters | Baseline, Days 14,,28,,42
  This was not a prespecified key secondary outcome
Vital signs | Baseline, Days ,14,21,28,42
  This was not a prespecified key secondary outcome
Weight | Baseline, Days 14,,28,,42
  This was not a prespecified key secondary outcome
Electrocardiograms (ECGs) | Baseline, Days ,14, 28, 42
  This was not a prespecified key secondary outcome
Adverse events (including serious adverse events) | Screen, baseline, Days 4,7,14,21,28,35,42 and recorded continuously for AEs up to 7 days after endpoint
  This was not a prespecified key secondary outcome
Serious adverse events (SAEs) up to 30 days after endpoint | Screen, baseline, Days 4,7,14,21,28,35,42 and recorded continuously for AEs up to 30 days after endpoint
  This was not a prespecified key secondary outcome

REFERENCES:
- [Result] Szegedi A, Verweij P, van Duijnhoven W, Mackle M, Cazorla P, Fennema H. Meta-analyses of the efficacy of asenapine for acute schizophrenia: comparisons with placebo and other antipsychotics. J Clin Psychiatry. 2012 Dec;73(12):1533-40. doi: 10.4088/JCP.11r07596. PMID 23290326